CLINICAL TRIAL: NCT02765958
Title: Analyze Sleep Stages by Portable ECG Device
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ping-Huai Wang, Chief, Far Eastern Memorial Hospital
Other Study IDs: FEMH-104181-F
Record Dates: First submitted 2016-05-04; First posted 2016-05-09 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy: subjects without heart disease or arrhythmia, no evidence of obstructive sleep apnea
  Interventions: Device: portable ECG devise
- OSA: obstructive sleep apnea
  Interventions: Device: portable ECG devise

INTERVENTIONS:
Device: portable ECG devise

SUMMARY:
Sleep is a fundamental need for human and is associated with the working performance and the disease occurrence. Furthermore, the amount of people with sleep disorder or apnea increased largely. Thus, the analysis of sleep stages and the measurement of sleep quality became more important recently. In clinical settings, the analysis of daily sleep quality depends on actigraphy and sleep log. However, the uses of actigraphy and sleep log are not really convenient for patients. In this trial, the investigators will measure the subjects' ECG signal and movement using a portable ECG device with motion sensor. On the other hand, the sleep stages are also obtained from the current wide-established measurement- polysomnography. The ECG signals, movements, and sleep stages will be analyzed by our algorithm of artificial neural network. Then, the investigators can obtain the preliminary analysis of sleep quality can be obtained by using ECG device with our algorithm. It is helpful for doctors to realize the patent's sleep quality quickly

ELIGIBILITY:
Inclusion Criteria:

* OSA: OPD OSA patients; Healthy: no OSA

Exclusion Criteria:

* heart disease
* arrhythmia

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient in chest clinic
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
RR interval changes compared to the report of polysomography | 8 hours
  The difference of RR interval in healthy subjects and obstructive sleep apnea subjects

CONTACTS AND LOCATIONS:
Overall Officials: Ping-huai Wang, MD, Principal Investigator — Far Eastern Memeorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes